CLINICAL TRIAL: NCT02642510
Title: Improving Patient Education for Newly Diagnosed Lymphoma and Acute Leukemia Inpatients
Brief Title: Improving Patient Education for Lymphoma and Leukemia Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Christina Peters, Advanced Practitioner, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00073387
Record Dates: First submitted 2015-12-27; First posted 2015-12-30 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DVD Structured Education (Experimental): Participants in this group will watch an educational DVD in addition to standard teaching by nursing staff.
  Interventions: Other: Structured Education DVD + Verbal Teaching; Other: Verbal Teaching
- Standard Educational Teaching (Active Comparator): Participants in this group will receive educational teaching by their assigned nursing staff.
  Interventions: Other: Verbal Teaching

INTERVENTIONS:
Other: Structured Education DVD + Verbal Teaching — The structured education DVD is a 15-minute DVD presentation of information about unit routines and activities; leukemia/lymphoma; treatment modalities and procedures; treatment of side effects; and participant and family members activities of importance to prevent infection and promote well-being during cancer treatment.
  Participants will also receive verbal educational teaching by their assigned nursing staff regarding information about leukemia and lymphoma, common treatments, and side effects.
  Arms: DVD Structured Education
Other: Verbal Teaching — Participants will receive verbal educational teaching by their assigned nursing staff regarding information about leukemia and lymphoma, common treatments, and side effects.

SUMMARY:
The purpose of this study is to evaluate the impact of a structured, DVD educational intervention about what to expect during inpatient treatment of a newly diagnosed cancer. The focus of the study will be newly diagnosed lymphoma and acute leukemia patients and their family members. Outcome variables will be the patient and family member's satisfaction with inpatient teaching and anxiety about inpatient treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of a structured, DVD educational intervention about what to expect during inpatient treatment of a newly diagnosed cancer. The focus of the study will be newly diagnosed lymphoma and acute leukemia patients and their family members. Outcome variables will be the patient and family member's satisfaction with inpatient teaching and anxiety about inpatient treatment.

The experimental group will watch a DVD educational presentation of information about unit routines and activities; leukemia/lymphoma; treatment modalities and procedures; treatment of side effects; and patient and family members activities of importance to prevent infection and promote well-being during cancer treatment.

Participants in the control group will receive usual educational teaching by their assigned nursing staff.

ELIGIBILITY:
Inclusion Criteria:

For participants admitted for suspect diagnosis of leukemia or lymphoma:

* Admission to the hematology/leukemia unit (6E) at Emory University Hospital with a suspected or actual new diagnosis of leukemia or lymphoma within the past 24 hours
* English-speaking
* Completed education to at least the 6th grade level
* No significant auditory or visual deficits with corrective devices
* No central nervous system involvement of disease
* Physiologically stable
* Not at end of life
* No alterations in mental status
* Agrees to family member (family member; significant other; friend) participation in study and to selecting the individual who could participate

For Family Members:

* Willing to view DVD and read education booklet
* Selected by patient to participate
* English speaking
* No significant auditory or visual deficits with corrective devices
* No alterations in mental status
* Completed education to at least the 6th grade level

Exclusion Criteria:

* At end of life
* Altered mental status
* Significant auditory or visual deficits with corrective devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-06; Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Quality of Discharge Teaching Scale (QDTS) Score | Post Educational Teaching (Up to 30 minutes)
  Overall satisfaction will be measured with the Quality of Discharge Teaching Scale (QDTS).The QDTS is a 24 item survey to evaluate all of the teaching received by patients during their hospitalization prior to discharge. Each item on the survey is rated on a 0 to 10 numeric scale, with 0 representing an item was not addressed and 10 representing an item addressed a great deal. For each aspect of education or information being evaluated, participant are asked to rate the content of the education, as well as the delivery of the content.

SECONDARY OUTCOMES:
Visual analog scale (VAS) Score | Post Educational Teaching (Up to 30 minutes)
  Participants are instructed to place a horizontal mark across the 100 mm vertical line anchored at one end with the words "No Anxiety" and at the other end "Worst Anxiety Imaginable" at the level of their anxiety about inpatient cancer treatment. Rating of anxiety for the study will be done by having the participant mark their anxiety level on a new, unmarked VAS. Scoring of the VAS is done by measuring in millimeters from the end of the vertical line with the anchor phrases of "no anxiety" to the intersection of the participant's mark on the vertical line. Possible scores on the VAS range from 0 to 100 millimeters with higher scores indicating higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Peters, NP, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States